CLINICAL TRIAL: NCT01580709
Title: Optimizing the Role of ERCP in Evaluating Indeterminate Bile Duct Strictures
Brief Title: Endoscopic Retrograde Cholangiopancreatography (ERCP) Based Sampling of Indeterminate Bile Duct Strictures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Gregory A. Cote, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 10895519; K23DK095148 (NIH)
Record Dates: First submitted 2012-04-17; First posted 2012-04-19 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Indeterminate Bile Duct Stricture
Keywords: stricture; cholangiocarcinoma; pancreatic adenocarcinoma; bile duct; ERCP
MeSH Terms: conditions — Constriction, Pathologic; Cholangiocarcinoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multimodality Approach (Active Comparator): Patients in the multimodality arm will undergo a single brushing for routine cytology, a second brush sample for Fluorescence In Situ Hybridization and a cholangioscopy with site-directed biopsies for histology.
  Interventions: Procedure: Multimodality tissue sampling
- Multiple brush samples (Active Comparator): In patients randomized to multiple brushing samples, subsequent brushings #2-7 will be labeled separately and consecutively and sent to cytology. The cytopathologist will review each specimen for cellularity using a previously validated scoring system and presence of malignancy (positive, highly suspicious, atypical, normal).
  Interventions: Procedure: Multiple brushings

INTERVENTIONS:
Procedure: Multiple brushings — Seven consecutive brush samples for cytology.
  Arms: Multiple brush samples
Procedure: Multimodality tissue sampling — Single brush for cytology + single brush for FISH + cholangioscopy with site-directed biopsies
  Arms: Multimodality Approach

SUMMARY:
Differentiating malignant from benign bile duct strictures is a conundrum, since no diagnostic test is highly sensitive for diagnosing cancer. While ERCP is effective in palliating obstructive jaundice, standard diagnostic tools in ERCP have a low diagnostic sensitivity and confirm the stricture's etiology in <50% of cases. During the first ERCP, standard practice is to obtain routine cytology (RC) using a single brush sample. If this is not diagnostic, patients often undergo repeat ERCP, endoscopic ultrasound or other, increasing health care costs. The incremental yield of performing alternate ERCP-based diagnostic tools during the first ERCP including fluorescence in situ hybridization (FISH), cholangioscopy w/biopsy and multiple brushes for routine cytology is currently unknown. There are no studies quantifying the amount of testing utilized to firmly diagnose the etiology of the stricture, or the most efficient combination of diagnostic tools during the first ERCP. These are important knowledge deficiencies since a definitive tissue diagnosis during the first ERCP could reduce the need for downstream tests and expedite treatment, thereby improving patient-centered and economic outcomes. The added costs of using multiple tools during the first ERCP may be offset by these benefits.

Among patients with indeterminate bile duct strictures, the investigators hypothesize that a multimodality approach will be more sensitive without a significant reduction in specificity compared to multiple brush samples for routine cytology. The investigators will test this hypothesis using an experimental trial design by randomizing patients during their first ERCP to multiple brushing samples for cytology vs. a single brush sample for cytology + FISH + cholangioscopy w/biopsy. To obtain preliminary data for a definitive multi-center trial, the investigators propose a pilot and feasibility study to compare the performance characteristics of each approach by evaluating the prospective clinical course, including treatment delay, quality of life, and life expectancy for each enrolled patient. If our hypothesis is validated in a subsequent definitive study, the standard approach to tissue sampling during the first ERCP may be altered.

ELIGIBILITY:
Inclusion Criteria:

* Extrahepatic BDS with no discrete mass on CT/MRI (either or both)
* A BDS is defined as a segmental narrowing of the bile duct > 50% of the proximal or distal unaffected duct.
* Biochemical evidence of cholestasis (increase in alkaline phosphatase ≥ 2x upper limit of normal ± total bilirubin ≥2.0mg/dL)

Exclusion Criteria:

* No clinical suspicion for malignancy
* Associated mass seen on CT or MRI
* Age ≤18, pregnancy, incarceration, inability to give informed consent
* Inability to undergo standard ERCP (e.g., postsurgical anatomy)
* Previous ERCP with sampling of BDS, other than a single brushing specimen sent for routine cytopathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Performance characteristics | 12 months
  A definite diagnosis of malignancy (i.e., "true positive") will be defined as either 1) a cytological or histological interpretation "positive for malignancy" based on brushing for RC or biopsy; 2) subsequent cytological or histological confirmation of malignancy within one year of the index procedure, via repeat ERCP, surgery, other diagnostic test.
  If a diagnosis of cancer is not confirmed after one year of follow-up, then the stricture will be classified as non-malignant and the negative cytology, FISH and histology from the index ERCP considered "true negatives."

SECONDARY OUTCOMES:
Incremental yield of multiple brushings | 12 months
  The additive role of each additional brushing will be analyzed for 1) adequacy of cellularity for cytological interpretation and 2) assessment of malignancy. The cytopathologist will be asked to interpret each of these outcomes using the first pass only (control group), first two passes only, first three passes only, and so on until all seven brushings are analyzed. The performance characteristics (see primary outcome) will be compared for each incremental brushing, assuming that a single intraductal brushing for RC is the reference standard.
Incremental cost effectiveness ratio | 12 months
  Complete data on medical utilization (e.g. hospitalizations, procedures, ambulatory visits) will be collected prospectively using Indiana Network for Patient Care (INPC) health information exchange databases (clinical electronic health record (EHR) and claims). Direct costs associated with the diagnostic evaluation of the indeterminate bile duct stricture (BDS) will be measured in both groups, including those costs associated with the index ERCP and all treatment costs associated with each study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Cote, MD, MS, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Medical University of South Carolina, Charleston, South Carolina